CLINICAL TRIAL: NCT07314762
Title: Elderly Patients Undergoing Surgery During Perioperative Period: a Prospective Cohort Study
Brief Title: Elderly Patients Undergoing Surgery During Perioperative Period
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Ting Li, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Other Study IDs: SAHoWMU-CR2025-03-231
Record Dates: First submitted 2025-12-11; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Complications; Elderly; Postoperative Delirium (POD); Risk Prediction Model; Pathogenesis
Keywords: postoperative delirium; elderly; Cohort study
MeSH Terms: conditions — Postoperative Complications; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid (CSF) samples (when available)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical patients aged 65 years or older: For the surgical group patients, questionnaires and scales measuring cognitive function, sleep quality, and quality of life were collected preoperatively, at 1-7 days post-operation, 30 days post-operation, and 1 year post-operation. During the operation, blood, cerebrospinal fluid, and other biological samples from the patients were also collected.
- non-surgical subjects aged 65 years or older: For the non-surgical group patients, patients' basic information was collected, along with cognitive scales, sleep scales, and quality of life questionnaires.

SUMMARY:
The elderly patients have poorer overall conditions and have lower tolerance to trauma, anesthesia, and surgery. Therefore, the incidence of postoperative complications is relatively higher. In non-cardiac surgeries, approximately 20% of elderly patients experience postoperative complications, and the incidence of postoperative delirium (POD) is 23.8%. This may lead to prolonged hospital stays, increased hospital costs, and affect prognosis and even mortality. The investigators plan to conduct a prospective cohort study by systematically collecting biological samples and clinical information of elderly patients during the perioperative period to explore the possible risk factors and pathogenesis of postoperative delirium and postoperative complications in elderly surgical patients, and to construct a risk prediction model for postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

1) Surgical patients aged 65 or above or non-surgical subjects aged 65 or above. 2) Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1）Refused to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Surgical patients aged 65 or above or non-surgical subjects aged 65 or above
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium (POD) within 7 days after surgery | Preoperative, postoperative day 1, 3, 5 and 7
  POD is diagnosed daily using the Three-Minute Diagnostic Confusion Assessment Method (3D-CAM).

SECONDARY OUTCOMES:
The types of postoperative delirium | Preoperative, postoperative day 1, 3, 5 and 7
  The type of delirium is assessed using the Richmond Agitation-Sedation Scale (RASS). The Richmond Agitation-Sedation Scale (RASS) is a 10-point scale ranging from -5 (unarousable) to +4 (combative). A score of +4 represents a combative state where the patient is violent and poses immediate danger, while a score of -5 indicates no response to any stimulus. Based on the RASS score, delirium can be categorized into three motoric subtypes: Hyperactive delirium: RASS scores consistently between +1 and +4. Hypoactive delirium: RASS scores consistently between 0 and -3. Mixed-type delirium: RASS scores that fluctuate between positive and negative values over the observation period.
The severity of postoperative delirium | Preoperative, postoperative day 1, 3, 5 and 7
  The severity of postoperative delirium will be assessed using the Confusion Assessment Method-Severity scale (CAM-S).
The duration of postoperative delirium | Preoperative, postoperative day 1, 3, 5 and 7
  Duration is defined as the number of days from the onset of delirium symptoms to symptom resolution or hospital discharge, whichever occurs first.
Postoperative neurocognitive dysfunction | Preoperative, postoperative day 1, 5, 30, and at 1 year.
  Neurocognitive decline is assessed by comparing baseline to postoperative scores on: Mini-Mental State Examination (MMSE, 0-30, higher=better function), Montreal Cognitive Assessment (MoCA, 0-30, higher=better function); and five neuropsychological tests-Clock Drawing Test, (DST, 0-16, higher=better attention), Trail Making Test Parts A and B (TMT-A/B, seconds, lower=better), Boston Naming Test (BNT, 0-30, higher=better naming), Auditory Verbal Learning Test - Huashan version (AVLT-H delayed recall, 0-10, higher=better memory), and Clock Drawing Test (CDT, 0-10, higher=better visuospatial/executive function). Patient/caregiver reports are also collected.
Hospital Anxiety and Depression Scale (HADS) score | Preoperative, postoperative day 1, 5, 30, and at 1 year.
  The Hospital Anxiety and Depression Scale (HADS) is used for assessment, with each subscale (anxiety or depression) scored from 0-21: "0-7: Non-case", "8-10: Doubtful case", "11-21: Definite case". Higher scores clearly indicate worse outcomes, i.e., more severe anxiety or depression symptoms.
Activity of Daily Living | Preoperative, postoperative day 1, 5, 30, and at 1 year.
  The Activities of Daily Living (ADL) are typically assessed using the Barthel Index. 0-100. A higher score indicates stronger independence: a score of 100 represents complete independence; a score of 61-99 suggests mild functional impairment with basic self-care ability; and a score of ≤40 indicates severe functional impairment, with significant or complete reliance on others for daily living.
Acute pain | Preoperative, postoperative day 1 and 3
  Using Visual Analogue Scale (VAS), 0-100, 0 means no pain, 100 means severe pain
Sleep quality | Preoperative, postoperative day 5, 30, and at 1 year.
  Sleep quality is assessed using the Pittsburgh Sleep Quality Index (PSQI). The total score ranges from 0 to 21 points. A score greater than 7 (>7) is typically considered the clinical cutoff for poor sleep quality. A higher score indicates poorer sleep quality.
Quality of Life Score | Preoperative, postoperative day 5, 30, and at 1 year.
  using EQ-5D(Score of EuroQol Five Dimensions Questionnaire (EQ-5D)) to measure quality of life
The FRAIL Scale | Preoperative, postoperative day 5, 30, and at 1 year.
  The FRAIL (Fatigue, Resistance, Ambulation, Illnesses, and Loss of Weight) Scale ranges from 0 to 5. A score of 0 indicates robust/non-frail status, scores of 1-2 indicate pre-frail status, and scores of 3-5 indicate frail status.
Length of hospitalization | till the day of discharge from hospital, an average of 7 days
  Length of hospital stay are measured from the anesthesia starting day to the discharge day
Mortality | During hospitalization, and postoperative day 30 and at 1 year.
  In-hospital mortality; 30-day postoperative mortality; 1-year postoperative mortality
Days at home up to 30 days after surgery (DAH30) | up to 30 days after surgery
Economic indicators | during the entire trial, an average of 1 year.
  Hospitalization fees; -Preoperative fees; -Anesthesia fees; -Surgery fees; -Post-operative fees; -Post-discharge medical expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Li, MD. PhD, Principal Investigator — Department of Anaesthesiology and Perioperative Medicine, The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication with no end date
Access Criteria: De-identified participant data underlying the findings will be made available upon reasonable request. Proposals for data access should be directed to the corresponding author (liting1021@aliyun.com).
URL: https://www.wzhealth.com/